CLINICAL TRIAL: NCT02233309
Title: Epidural Pressure Changes Following Caudal Blockade: A Prospective Observational Study
Brief Title: A Prospective Observational Study of Epidural Pressures During Caudal Epidural in the Pediatric Population
Status: Completed | Type: Observational
Sponsor: Jessica Goeller (Other)
Responsible Party: Sponsor-Investigator, Jessica Goeller, Anesthesiology Fellow, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: IRB14-00119
Record Dates: First submitted 2014-08-01; First posted 2014-09-08 (Estimated); Results first posted 2015-05-28 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Anesthesia, Caudal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Monitoring of pressures during caudal anesthesia: Patients receiving caudal anesthesia as standard of care for a surgical procedure.
  Our study adds a monitoring line to the needle for the caudal. The caudal itself is not part of the study.
  Interventions: Other: Monitoring of pressures during caudal anesthesia

INTERVENTIONS:
Other: Monitoring of pressures during caudal anesthesia — The caudal itself is a separate procedure not covered by this observational study. This study simply attaches a monitoring device to the needle used for the caudal to measure pressures. The caudal takes place whether the observation of pressures is agreed to or not, as per standard protocol.

SUMMARY:
This study is a prospective study of epidural pressure changes when local anesthetic is injected from the caudal route. All patients will receive the same weight based volume dose of local anesthetic after induction of general anesthesia, and a CVP transducer will be attached to the standard caudal needle for measurement of pressure: under the skin, after entering the epidural space, and every 15 seconds for 3 minutes after completion of injection with the needle in situ. The placement of the caudal epidural will follow current standard of care and administration, the only variation will be the addition of a pressure transducer to the stopcock where the local anesthetic syringe is attached that will allow for pressure monitoring.

DETAILED DESCRIPTION:
After approval of the Internal Review Board, the patients and families will be given the opportunity to participate in the proposed research study if inclusion criteria are met. The patient/family will sign the anesthesia consent form, as per protocol, by initialing the box at the bottom that states 'I do want, if indicated, regional anesthetic techniques employed for anesthetic maintenance and/or port operative pain relief for my child.' The primary anesthesia team (anesthesiologist/CNRA/resident) will be made aware that the need for a pressure transducer for the caudal epidural injection will be required and that a member of the research team will be documenting pressures during the procedure. Premedication with midazolam will be at the discretion of the attending anesthesiologist covering the case. Anesthesia induction may be performed with either intravenous medications or mask inhalation at the attending anesthesiologist's discretion; however no narcotics will be administered during induction, as is common when a caudal epidural is utilized for post-operative pain control. The airway will be secured using an oral endotracheal tube or laryngeal mask airway (LMA).

The single shot caudal epidural block with pressure monitoring will be performed by one of the study investigators. Ropivicaine/Bupivacaine 0.125-0.25% will be used as the local anesthetic for the caudal epidural with a total dose not to exceed 1 ml/kg. Pressure transduction will be constantly in place, with pressures being recorded by a research nurse: 1) prior to entering the epidural space, but after needle introduction under the skin, 2) after loss of resistance upon entering the epidural space, 3) at 5 second intervals during injection of the 1 mL/kg bolus of local anesthetic 4) continuing with pressure monitoring for an additional minute, in 10 second increments, after the injection is completed. Following placement of the block, a band-aidwill be placed, where appropriate, and the patient will be prepped for the surgical procedure. The primary anesthesia team will continue delivering the general anesthetic for the remainder of the case. Maintenance anesthesia will be carried out per our usual routine.

Upon completion of the surgical procedure, the patient's airway device will be removed and the patient will be transferred to the post-anesthesia care unit (PACU). In the PACU, the principal or co-investigator will review the patient's treatment needs for pain in the PACU to determine whether the block was efficacious; fentanyl 0.5 µg/kg, or the morphine-equivalent dose, will be administered as necessary based on the pain assessment. The patients will be discharged from PACU when discharge criteria are met per the Aldrete score.

ELIGIBILITY:
Inclusion Criteria:

1. ASA physical status I or II
2. Weight ≥ 3 kilograms
3. Undergoing a lower abdominal/pelvic or urologic procedure where caudal epidural anesthesia is a beneficial adjunct

Exclusion Criteria:

1. Co-morbid diseases (cardiac, pulmonary, neurological disease)
2. Patients with sacral deformities contraindicating a caudal epidural
3. Use of therapeutic dose anticoagulants or presence of a bleeding disorder
4. Other co-existing conditions would preclude the use of neuraxial blockade

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who will be receiving caudal anesthesia as part of their surgical procedure.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2014-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Goeller, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Monitoring of Pressures During Caudal Anesthesia: Patients receiving caudal anesthesia as standard of care for a surgical procedure.
  Our study adds a monitoring line to the needle for the caudal. The caudal itself is not part of the study.
  Monitoring of pressures during caudal anesthesia: The caudal itself is a separate procedure not covered by this observational study. This study simply attaches a monitoring device to the needle used for the caudal to measure pressures. The caudal takes place whether the observation of pressures is agreed to or not, as per standard protocol.
Period: Overall Study
Arm/Group | Monitoring of Pressures During Caudal Anesthesia
Started | 36
Completed | 31
Not Completed | 5
Not completed — Physician Decision | 5

BASELINE CHARACTERISTICS:
Arm/Group | Monitoring of Pressures During Caudal Anesthesia
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 36
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 2.21 (2.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 36
Region of Enrollment [Number; unit: participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Pressure in the Caudal Epidural Space
Description: After administration of the single-shot bolus dose of the local anesthetic agent (1 mL/kg), the immediate post-bolus pressure was measured.
Time Frame: Immediately post bolus
Population: Due to errors in data collection or protocol violations, 5 patients were excluded leaving 31 patients for analysis.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Monitoring of Pressures During Caudal Anesthesia
Number analyzed (Participants) | 31
mmHg | 192.5 (93.3)

ADVERSE EVENTS:
Arm/Group | Monitoring of Pressures During Caudal Anesthesia
Serious Adverse Events (participants affected / at risk) | 0/36
Other Adverse Events (participants affected / at risk) | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes